CLINICAL TRIAL: NCT02237612
Title: Diffusion-Weighted MRI for Staging in Localized Prostate Cancer: A Pilot Study
Brief Title: Diffusion-Weighted MRI in Staging Patients With Localized Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4P-08-4; NCI-2014-01848 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-08-00413-CR004; HS-08-00413; 4P-08-4 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2014-09-04; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Adenocarcinoma of the Prostate; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (diffusion-weighted MRI) (Experimental): Patients undergo diffusion-weighted MRI of the pelvis.
  Interventions: Procedure: diffusion-weighted magnetic resonance imaging; Other: laboratory biomarker analysis

INTERVENTIONS:
Procedure: diffusion-weighted magnetic resonance imaging — Undergo diffusion-weighted MRI
  Other Names: diffusion-weighted MRI
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies how well diffusion-weighted magnetic resonance imaging (MRI) works in staging patients with prostate cancer that has not spread to nearby lymph nodes or other parts of the body. New imaging techniques, such as diffusion-weighted MRI, may be a less invasive way of predicting the stage and grade of prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the sensitivity and specificity of diffusion-weighted MRI for pathologic T3 stage prostate cancer using a 3 Tesla (3T) magnet with a surface coil.

OUTLINE:

Patients undergo diffusion-weighted MRI of the pelvis.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-documented adenocarcinoma of the prostate which is intermediate or high risk, defined as possessing one or more of the following features:

  * Gleason >= 7
  * > 50% biopsy cores +
  * Prostate-specific antigen (PSA) >= 10
* Interested in undergoing a radical prostatectomy as definitive management for prostate cancer
* No clinical or radiographic evidence for distant metastatic disease

  * In subjects with PSA < 20 no radiographic staging is required in the absence of clinical symptoms for distant metastatic disease; for those with PSA > 20, a bone scan must document lack of concern for bone involvement

Exclusion Criteria:

* Ineligible for surgery due to cardiac, pulmonary, or other major comorbidity factor
* History of claustrophobia
* Pacemaker or other implanted metal objects which would make subject ineligible for MRI, per standard criteria
* Unable to give written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of patients found to have extracapsular extension and seminal vesicle involvement using Diffusion-Weighted MRI | Baseline
  Patients will be imaged using diffusion-weighted MR. Findings will be correlated with histopathologic findings at biopsy and/or prostatectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Dorff, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States